

Official Title: PROTOCOL #: 7027-MCPL-2021

# HISTOLOGICAL STUDY TO ASSESS SAFETY AND EFFICACY OF THE TEMPSURE® FIRM FOR NON-INVASIVE LIPOLYSIS

NCT Number: NCT04878172 DOCUMENT DATE: MARCH 5, 2021



## INVESTIGATIONAL PLAN

## PROTOCOL #: 7027-MCPL-2021

## HISTOLOGICAL STUDY TO ASSESS SAFETY AND EFFICACY OF THE TEMPSURE® FIRM FOR NON-INVASIVE LIPOLYSIS

#### CONFIDENTIAL

THIS INVESTIGATIONAL PLAN CONTAINS CONFIDENTIAL INFORMATION FOR USE BY THE INVESTIGATORS AND THEIR DISIGNATED REPRESENTITIVES PARTICIPATING IN THIS STUDY. IT SHOULD BE HELD CONFIDENTIAL AND MAINTAINED IN A SECURE LOCATION. IT SHOULD NOT BE COPIED OR MADE AVAILABLE FOR REVIEW BY ANY UNAUTHORIZED ENTITY.

## **SPONSOR:**

CYNOSURE, LLC 5 CARLISLE ROAD WESTFORD, MA 01886 PHONE: 800-886-2966 FAX: 978-256-6556



## HISTOLOGICAL STUDY TO ASSESS SAFETY AND EFFICACY OF THE TEMPSURE® FIRM FOR NON-INVASIVE LIPOLYSIS

#### INVESTIGATOR AGREEMENT

I agree to conduct the study in accordance with the relevant, current protocol and will only make changes in a protocol after notifying the sponsor, except when necessary to protect the safety, rights, or welfare of subjects.

I agree to personally conduct or supervise the described investigation.

I agree to inform any patients, or any persons used as controls if applicable, that the device(s) is/are being used for investigational purposes and I will ensure that the requirements relating to obtaining informed consent in and institutional review board (IRB) review and approval are met.

I agree to report to the sponsor adverse experiences that occur in the course of the investigations. I have read and understand the information in the device manual, including the potential risks and side effects of the device.

I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed about their obligations in meeting the above commitments.

I agree to maintain adequate and accurate records and to make those records available for inspection. I further agree that Cynosure, Inc. or their designees shall have access to any source documents from which case report form information may have been generated.

I will ensure that an IRB that complies with the requirements of 21 CFR Part 56 will be responsible for the initial and continuing review and approval of the clinical investigation. I also agree to promptly report to the IRB all changes in the research activity and all unanticipated problems involving risks to human subjects or others. Additionally, I will not make any changes in the research without IRB approval, except where necessary to eliminate apparent immediate hazards to human subjects.

I agree to comply with all other requirements regarding the obligations of clinical investigators.

I will comply with the International Conference on Harmonization (ICH), Good Clinical Practice (GCP) guidance E6, FDA Good Clinical Practice Regulations (21 CFR parts 50, 56, and 812), Declaration of Helsinki (DoH) and the Health Human Service (HHS) Belmont Study Principals and Guidelines during the conduct of this study.

I have read the foregoing protocol and agree that it contains all necessary details for carrying out this study. I will conduct the study as outlined herein and will complete the study within the time designated.

I will provide copies of the protocol and all pertinent information to all individuals responsible to me who assist in the conduct of this study. I will discuss this material with them to ensure they are fully informed regarding the study device the conduct of the study.

I will disclose financial arrangements and interests in accordance with Financial Disclosure Rules (21 CFR part 54) and FDA Form 3455.

Investigator's Signature

Name of Investigator (Typed or Printed)

Address of Investigator (Typed or Printed)



## SITE #1 CONTACT INFORMATION:

## **Principal Investigator Information:**

Lawrence Bass, M.D Bass Plastic Surgery PLLC 568 Park Avenue New York, NY 10065 Phone: 212-593-2600

Email: <u>DrBass@DrBass.net</u>

## SITE #2 CONTACT INFORMATION:

## **Principal Investigator Information:**

John W. Decorato. M.D Aesthetic Pavilion Ambulatory Surgery Center 531 W 2777 Hylan Blvd Staten Island, NY 10306 Phone: 718-987-0300 Email: jwd@DrDecorato.com

## SITE #3 CONTACT INFORMATION:

## **Principal Investigator Information:**

Barry DiBernardo, M.D New Jersey Plastic Surgery 29 Park Street Montclair, NJ 07042 Phone: 973, 509, 2000

Phone: 973-509-2000 Email: <u>drd@njpsmd.com</u>

## SPONSOR CONTACT INFORMATION:

Jennifer Civiok Director, Clinical Development 5 Carlisle Road Westford, MA 01886 Phone: 978-399-4343

Email: Jennifer.Civiok@cynosure.com

David Canavan Sr. Clinical Project Manager Westford, MA 01886 Phone: 978-551-5786

Email: David.Canavan@cynosure.com



## TABLE OF CONTENTS

- 1.0 PURPOSE
  - 1.1 Name and Intended Use
  - 1.2 Objectives
  - 1.3 Duration of the Investigation
- 2.0 PROTOCOL
  - 2.1 Protocol Methodology and Analysis
  - 2.2 Protocol Study Design
  - 2.3 Subject Selection Criteria
  - 2.4 Screening
  - 2.5 Informed Consent Process and Enrollment
  - 2.6 Pre-Treatment Procedures
  - 2.7 Treatment Procedures
  - 2.8 Post Treatment Procedures
  - 2.9 Biopsy Portion of Study
  - 2.10 Follow Up
  - 2.11 Unscheduled Visits
  - 2.12 Replacement of Subjects
  - 2.13 Schedule of Visits and Procedures
  - 2.14 Evaluation Methods
  - 2.15 Adverse Event Recording
  - 2.16 Statistical Analysis
- 3.0 RISK ANALYSIS AND MANAGEMENT
- 4.0 DEVICE DESCRIPTION AND SPECIFICATIONS
- 5.0 MONITORING PROCEDURES
- 6.0 LABELING
- 7.0 CONSENT MATERIALS
- 8.0 INSTITUTIONAL REVIEW BOARD INFORMATION
- 9.0 OTHER INSTITUTIONS
- 10.0 ADDITIONAL RECORDS AND REPORTS
- 11.0 PREGNANCY
- 12.0 SUBJECT WITHDRAWAL
- 13.0 PHOTOGRAPHY
- 14.0 ADVERSE REACTIONS DEFINITIONS AND REPORTING REQUIREMENTS
- 15.0 PROTOCOL DEVIATIONS
- 16.0 CONFIDENTIALITY AND DISCLOSURE OF MEDICAL INFORMATION
- 17.0 CLINICAL RESEARCH CONDUCT
- 18.0 REPORTING FOR THE STUDY
- 19.0 DISCLOSURE
- 20.0 RESPONSIBILITY OF THE INVESTIGATOR
- 21.0 PROCEDURE FOR AMMENDMENTS TO PROTOCOL
- 22.0 TERMINATION OF STUDY
- 23.0 DATA SECURITY
- 24.0 REPORT OF PRIOR INVESTIGATIONS

## **APPENDICES**

- A. Protocol Revisions Tracker
- B. Universal Pain Assessment Tool



## ATTACHMENTS/REFERENCES

- I.
- Operator Manual for the TempSure® Clinical Reference Guide for the TempSure® II.
- III. Informed Consent Form
- IV. Pre and Post Treatment Instructions
- V. Advertisement (optional)



#### **PURPOSE**

### 1.1 Name and Intended Use

The device used in this study is called TempSure®.

The intended use of the TempSure® device is to use the Firm handpieces for non-invasive lipolysis.

## 1.1 Objectives

- 1. Primary Objectives:
  - To demonstrate adipocyte injury confirmed by histology.
- 2. Additional Assessment:
  - Ultrasound measurements. (optional)
  - Evaluation of thermal imaging taken of the treatment during device use. (optional)
  - Safety assessment through the collection of Adverse Events.

#### 1.2 Duration of the Investigation

The sponsor anticipates that all subjects can be enrolled within 3 months. If subject participates in all visits, then the subject's participation in this study may last up to 2 months. It is anticipated that it will take approximately 3 months to analyze the data collected during this study. The total duration of this study is anticipated to last approximately 8 months.

#### 2.0 PROTOCOL

## 2.1 Protocol Methodology and Analysis

#### Methodology:

Subjects are to be enrolled in this clinical study if they are 18-55 years old and are willing to have biopsies taken from a control site and the treatment area. Subjects may be enrolled if they have been previously scheduled or are willing to have an abdominoplasty procedure at one of the study specified timepoints, after being treated with the study device . A maximum of 12 subjects will be enrolled at up to 3 study centers. Subjects will attend a screening/pretreatment visit which may be performed on the same day as the treatment visit. Subjects may receive 1 treatment with the TempSure® Firm on the abdomen. Subjects may receive a phone call 1 week (1-10 days) post each treatment. Subjects will undergo abdominoplasty surgery at one of four predetermined timepoints after an abdomen treatment with TempSure® Firm: day 0 (within 24 hours after treatment), 10 days (+/- 3 days), 20 days (+/- 3 days), or 30 days (+/- 7 days). This will be determined on availability of the subject and/or on an as needed basis and this will be decided by the investigator and Sponsor. An unscheduled visit or phone call may be performed at any time during the study at the subject's request or as deemed necessary by the site Investigator.

## Analysis:

Upcoming generations are proving to have an interest in non-ablative aesthetic treatments and will drive demand for innovated products, procedures, and practice design. Due to this shift in patient base, practices need to evolve to adapt to the newer generational ideologies. There have been rapid advances in RF technology over the past few years and the nonsurgical treatment using this energy source offers great promise to our aging population. Radiofrequency technology for lipolysis needs to be further investigated to optimize treatment parameters for safe and effective non-ablative aesthetic treatments.

#### Relevance:

Non-invasive fat reduction is a commonly sought out procedure and continues to increase in demand (+3% from 2018 to 2019)<sup>3</sup> perhaps because, according to the CDC, the prevalence of obesity in the U.S. was 42.4% in 2017-2018<sup>4</sup>. Currently, the treatments available for non-invasive lipolysis include, but not limited to, radiofrequency, cryolipolysis, laser lipolysis, HIFEM, and ultrasound. The limitations of current products on the market include different side effect profiles and modes of administration.

#### Testability:

The truSculpt device has been cleared for used using the 2 MHz setting for the 40cm<sup>2</sup> handpiece for reduction in circumference of the abdomen and non-invasive lipolysis of the abdomen (FDA K180709). The truSculpt study



\_\_\_\_\_\_

utilized the collection of biopsies and safety data. This study will utilize the histology data from multiple biopsies collected at specified timepoints and safety data to evaluate the safety and efficacy of the treatment.

## Compatibility:

Due to such a high prevalence of obesity in the U.S. and the increasing demand for non-invasive lipolysis treatments, there is a need to treat unwanted fat in its earlier stages to optimize treatment outcomes. As a subject gets older or the condition worsens, treatments may need to be more aggressive to get the same response as younger subjects or less severe cases.

#### Predictive power:

While this study will observe lipolysis effects of treatments with TempSure® handpieces on the abdomen, results could potentially be applied to a variety of body areas..

## 2.2 Protocol Study Design

This is a prospective, open-labeled, non-randomized, multi-center clinical study to collect safety and efficacy data on the TempSure® Firm.

## 2.3 Subject Selection Criteria

Subjects will meet the criteria described below:

#### Inclusion Criteria:

- Male or female between 18 55 years old.
- Willing to receive treatments with the TempSure® device and willing to have biopsies taken from a control site and the treatment area (biopsies are collected after the abdominal tissue flap is removed during abdominoplasty surgery)
- Understand and accept obligation not to receive any other procedures on the treatment and control areas throughout the length of the study.
- Understand and accept the obligation and able to be present for all study visits
- Willing to comply with all requirements of the study and able to provide informed consent.

#### **Exclusion Criteria:**

- Pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning to become pregnant prior to the end of the study.
- Currently enrolled in an investigational drug or device trial, or has received an investigational drug or investigational device treatment(s) in the area to be treated (or designated control area) 6 months prior to entering this study (or at the discretion of the Investigator).
- Cuts, wounds, or infected skin on the area to be treated or designated control area
- On local, oral, or systemic anesthetic agents.
- Condition(s) or circumstance(s) that, in the investigators opinion, may put the subject at significant risk, may confound study results or may interfere significantly with subject participation.

## Cautionary Criteria:

- Any embedded electronic device that gives or receives a signal, the device should be turned off or removed prior to treatment.
- Embedded pacemaker or implantable cardioverter defibrillator (ICD), the client's cardiologist must be consulted prior to treatment.
  - **NOTE**: This device has not been tested on patients implanted with electronic devices that receive or emit signals, such as: Pacemakers, Implantable Cardiac Defibrillators (ICD), or Cardiac Resynchronization Therapy (CRT) devices.
- If the neutral pad would need to be placed on a subject that has a metal plate, rod, or any metal implant that could conduct heat from the Smart Handpiece or surgical handpiece.
- Allergy to adhesives, such as glues on medical tape, they should be alerted that a rash may occur on the neutral pad site and an over-the-counter solution may be used to treat the area.
- Allergy to gold, such as the metallic covering of the TempSure handpieces.



- Allergy to corn, such as the corn derivative ingredient in Parker Aquasonic Gel.
- If the subject has an unhealthy expectation of the results treatment with the TempSure device is not plastic surgery; all subjects should be fully informed of the expected treatment results.
- Nerve insensitivity to heat in the treatment area.
- Severe laxity or sagging that causes redundant folds of tissue or hanging skin in the area to be treated this treatment will be ineffective.
- Accutane (Isotretinoin) use six to twelve months prior to treatment, as this can thin the skin and make it brittle.
- Studies of the use of the RF generator on subjects that have any of the following conditions is unknown:
  - Autoimmune Disease
  - Diabetes
  - Herpes Simplex
- Use caution when treating areas that have scars, tattoos, permanent makeup, and permanent brows.

List any concomitant medications or procedures permitted before, during and after the trial.

Subjects will be recruited for the study through investigator's existing patient databases and advertisements.

Subject populations will not be eligible to participate in the study if they are vulnerable populations such as children, pregnant women, prisoners, institutionalized individuals, and any persons requiring a legally authorized representative as part of the consenting process.

Subject population characteristics that will not be eligible to participate in the study include non-English speaking individuals and people who cannot read or comprehend English.

#### 2.4 Screening

Subjects will be asked questions about their medical history, inclusion/exclusion criteria will be verified, and a limited physical exam may be performed. If applicable, discontinuation of concomitant medications will be discussed with subject. Pre and post treatment instructions will be reviewed with the subject. Subjects will be informed of standard COVID-19 procedures that adhere to federal and state guidelines.

## Procedure for the Limited Physical Exam:

If the investigator determines a limited physical exam is necessary, the exam will be similar to a basic annual physical exam performed by a qualified clinician to determine general overall health. The limited medical exam may include any or all of the following; vital signs such as blood pressure, heart rate, respiratory rate and body temperature, general appearance, listening to the heart, lungs and abdomen with a stethoscope, head and neck exam, in addition to examining the throat, tonsils, teeth, ears, eyes and nose as well as a neurological exam such as testing muscle strength, reflexes, balance and mental state.

The following pre-treatment instructions will be reviewed:

- Shave any dense hair on the area to be treated.
- Do not wear constrictive clothing. Treatment area must be accessible. The back for the neutral pad will also need to be accessed.
- o Treatment and control areas must be free of any cuts, scratches, open lesions or infection.
- For optimum treatment, hydrate by drinking water (at least 8 cups daily) or hydrating fluids such as Gatorade.
   Avoid drinking alcohol for 24 hours in advance.

The following post treatment instructions will be reviewed:

- o If the skin is slightly pink or red in areas following the treatment, avoid hot water when washing or showering until any erythema (redness) has subsided.
- o Soothing creams or moisturizers, such as Aveeno, may be used.
- o Gently massage the treated area daily for 5 minutes for the duration of your involvement in the study.
- o Use a sun block with UVA and UVB protection with SPF of 30 or greater to prevent sun damage.
- o Maintain the same weight and exercise routine throughout the study.



## 2.5 Informed Consent Process and Enrollment

Subjects will be asked to review the pre and post treatment instructions prior to signing the informed consent form and prior to involvement in the study. Subjects who sign the informed consent will be screened to confirm eligibility and, if eligible, will be assigned a subject identification number. Subjects will be de-identified through their subject identification number, which will be stored in a secure location. Subject identification numbers will be generated chronologically and assigned only to subjects who have met all the study selection criteria and have signed the informed consent form. Informed consent will be obtained prior to a subject's involvement in study related procedures. A subject will be considered enrolled in the study once they have signed the informed consent form.

## 2.6 Pre-Treatment Procedures

If the subject is of childbearing potential (i.e., females not post-menopausal or not surgically sterile), they will be asked if they are pregnant and date of last menstrual cycle. Prior to treatment, a urine pregnancy test will be performed on all women of childbearing potential. A urine pregnancy test may also be conducted at the Investigator's discretion at any time during the study. If a urine pregnancy test is conducted, a negative result must be obtained within 24 hours prior to the treatment.

## Urine Pregnancy Test Procedure:

- o A urine sample is tested mid-stream or by cup sample with an indicator stick.
- o Negative results are indicated on the indicator stick.
- The area to be treated will be identified and may be marked with a surgical marker.
- Photographs will be taken prior to and after the treatment(s).
- An ultrasound will be performed prior to the treatment.
- The treatment area and the neutral pad area may be cleansed with water and soap and/or alcohol.
- The neutral pad will be placed on the back in an area determined by the Investigator to optimize and maintain device energy settings during the treatment.

## **2.7 Treatment Procedures**

- The Investigator will use the device as described in the TempSure Operator's Manual and Clinical Reference Guide.
- Gel will be applied to the treatment area.
- The TempSure® Firm handpiece (25mm, 30mm, 60mm) to be used and the limits of the area to be treated will be determined by the Investigator and may be used in accordance with the TempSure Clinical Reference Guide.
- The handpiece will be placed in contact with the skin.
- The entire defined treatment area will be treated by delivering energy to the skin.
- Parameters may be adjusted throughout the treatment to increase subject comfort.
- Subjects will be asked to report the general level of treatment discomfort/pain on a scale of 0 (none) to 10 (maximum intolerable pain).
- Temperature will be continuously monitor using thermal imaging and recorded during treatment.
- Photographs may be taken at any time during treatment to document treatment area and, if applicable, any adverse
  events.

## **2.8 Post Treatment Procedures**

- Adverse events will be documented after treatment.
- Post treatment instructions will be reviewed.
- Photographs may be taken.
- Ultrasounds may be performed

## 2.9 Biopsy Portion of the Study

- Subjects must be scheduled for abdominoplasty surgery, up to 20 biopsies may be taken from the abdominal tissue that is removed at the time of surgery.
- Biopsies will be taken from treatment and control sites



## 2.10 Follow Up

- Subjects may receive a phone call 1 week (1-10 days) after treatment(s) to record observations and/or side effects.
- Subjects may return for follow up visit at 10 days, 20 days, and/or 30 days after the treatment.
- Biopsies will be taken on a predetermined date of abdominoplasty surgery.
- Photographs and ultrasounds may be taken at all follow up and unscheduled visits.
- Adverse events will be documented at all follow up and unscheduled visits.

## 2.11 Unscheduled Visits

An unscheduled visit may be performed at any time during the study at the subject's request or as deemed necessary by the site Investigator. The date and reason for the unscheduled visit will be recorded in the source documentation.

## 2.12 Replacement of Subjects

Replacement of subjects who have withdrawn or been withdrawn from the study will be allowed to be replaced with prior approval from the sponsor and.



## 2.13 Schedule of Visits and Procedures

Day 0 Biopsy Group

| Day o Biopsy Group | | |
|---|---|---|
| | Visit #1* | Visit #2 |
| Procedure | Screening<br>and<br>Pre-<br>treatment<br>Procedures | Treatment<br>Visit |
| Medical History | X | |
| Pregnancy Verification** | X | X |
| Informed Consent | X | |
| Photographs | X | X |
| Ultrasound | X | X |
| Treatment | | X |
| Treatment Discomfort/ Pain Evaluation | | X |
| Adverse Events<br>Assessment | X | X |
| Abdominoplasty and Biopsies | | X |

Day 10 Biopsy group

| | Visit #1* | Visit #2 | Call | Visit #3 |
|---|---|---|---|---|
| Procedure | Screening<br>and<br>Pre-<br>treatment<br>Procedures | Treatment<br>Visit | Phone Call<br>1 Week<br>Post Tx<br>(1-10 Days) | 10 Days Follow<br>up<br>Post Tx<br>(+/- 3 Days) &<br>Abdominoplasty |
| Medical History | X | | | |
| Pregnancy Verification** | X | X | | |
| Informed Consent | X | | | |
| Photographs | X | X | | X |
| Ultrasound | X | X | | X |
| Treatment | | X | | |
| Treatment Discomfort/ Pain Evaluation | | X | | |
| Adverse Events<br>Assessment | X | X | X | X |
| Abdominoplasty and Biopsies | | | | X |



Day 20 Biopsy group

| Day 20 Diopsy group | | | | |
|---|---|---|---|---|
| | Visit #1* | Visit #2 | Call | Visit #3 |
| Procedure | Screening<br>and<br>Pre-<br>treatment<br>Procedures | Treatment<br>Visit | Phone Call 1 Week Post Tx (1-10 Days) | 20 Days Follow<br>up<br>Post Tx<br>(+/- 3 Days) &<br>Abdominoplasty |
| Medical History | X | | | |
| Pregnancy Verification** | X | X | | |
| Informed Consent | X | | | |
| Photographs | X | X | | X |
| Ultrasound | X | X | | X |
| Treatment | | X | | |
| Treatment Discomfort/ Pain Evaluation | | X | | |
| Adverse Events<br>Assessment | X | X | X | X |
| Abdominoplasty and Biopsies | | | | X |

Day 30 Biopsy group

| | Visit #1* | Visit #2 | Call | Visit #3 |
|---|---|---|---|---|
| Procedure | Screening<br>and<br>Pre-<br>treatment<br>Procedures | Treatment<br>Visit | Phone Call<br>1 Week<br>Post Tx<br>(1-10 Days) | 30 Days Follow<br>up<br>Post Tx<br>(+/- 7 Days) &<br>Abdominoplasty |
| Medical History | X | | | |
| Pregnancy Verification** | X | X | | |
| Informed Consent | X | | | |
| Photographs | X | X | | X |
| Ultrasound | X | X | | X |
| Treatment | | X | | |
| Treatment Discomfort/ Pain Evaluation | | X | | |
| Adverse Events<br>Assessment | X | X | X | X |
| Abdominoplasty and Biopsies | | | | X |

<sup>\*</sup>Screening and Pre-treatment Procedures may occur at the same time as the Treatment Visit .

<sup>\*\*</sup>Pregnancy verification required before each treatment only for women of childbearing potential.



## 2.14 Evaluation Methods

#### **Photographs:**

Photographs may be taken at all visits and will be used to assess safety of treatment.

## **Histology of Biopsy**

Biopsies of the excised tissue will be obtained and prepared for histology to examine the tissue response following RF treatment. Each specimen will first be preserved with a fixative and stained with Hematoxylin and eosin (H&E stain). Samples will be assessed independently and may be assessed for normal structures, cell viability, vascular injury, and overall morphologic traits, injury, and any indications of the healing response. A report will be provided to summarize finding for all samples.

## Ultrasound (U/S)

An ultrasound scan is a noninvasive diagnostic test that uses sound waves to capture live internal anatomical images of the body. Subjects will be lying down on a table with a section of the body exposed for the test. A special lubricating gel will be applied to the skin. This prevents friction between the ultrasound transducer—similar in appearance to a microphone— and the skin. The lubricating gel also helps transmit the sound waves during the scan. After the ultrasound e is performed, the gel will be cleaned off the subject with water. The ultrasound typically lasts less than 30 minutes.

## **Treatment Discomfort/Pain Evaluation:**

Subjects will be asked to report the general level of treatment discomfort on a scale of 0 (none) to 10 (maximum intolerable pain) using the universal pain assessment tool (Appendix B)

#### **Temperature Monitoring**

An infrared thermometer may also be used for temperature monitoring to measure temperature on the skin before, during, and after a treatment.

#### 2.15 Adverse Event Recording

All data captured must be supported by the Investigator's timely assessment and documentation of the adverse event in the case report forms or source documents. All documented adverse events will be reviewed by the Sponsor or designee to determine whether the adverse event meets regulatory reporting requirements and to ensure timely adverse event reporting in compliance with local and global regulatory requirements.

## Adverse Events Pertaining to the TempSure® Device:

Mild discomfort during treatment may be experienced by the subject. Typically, the discomfort is temporary and localized within the treatment area. Mild edema (swelling) and erythema (redness) may occur. Initial studies indicate that these side effects typically resolve within 2 to 24 hours.

Other anticipated side effects may include pain, skin burns, blistering, bleeding, scarring, crusting, bruising, infection, itching, prolonged edema (swelling) and erythema (redness), hardness, and nodules. Loss of hair pigment may also occur within and adjacent to the treatment area.

## **Adverse Events Pertaining to Ultrasound Gel:**

The gel is a water-based gel that may be placed on the skin during the TempSure® Firm treatment. No known adverse events are documented. However, an allergic reaction is always possible when placing a topical gel on the skin. Allergic reaction may include a mild reaction such as skin redness, irritation, or hives, all are typically transient and fully resolve.

## Adverse Events Pertaining to Neutral Pad:

Subject may feel mild heat or hot spots during the treatment(s). If the subject reports heat at the pad site, evaluate the site, check for epidermal injury. Skins burns may occur if subject does not report feeling excessive heat at the site of the pad.

## **Adverse Events Pertaining to Ultrasound:**

Ultrasound imaging has minimal risks and may produce effects on the body such as redness and pockets of gas. Skin rashes from use of the ultrasound gel may also occur.



## **Adverse Events Pertaining to the Surgical Marker:**

Using surgical marker has minimal risks and may produce effects on the body such as redness or a rash. Markings may remain visible for a few days or may be removed with mild soap or alcohol.

#### **Other Cautions:**

Incomplete response or no response may occur since some subjects may not respond to treatment.

## 2.16 Statistical Analysis

## 2.16.1 Hypothesis

For this study to be considered a success, biopsies from the from the treatment areas show adipocyte injury and/or inflammatory immune cell response to the subcutaneous fat.

## 2.16.2 Sample Size Rationale

Based on the need for repetition of results and comparison to predicate devices, it was determined that a total of 12 subjects will be required for this study.

#### 2.16.3 Patient Populations

Interim results may be collected and reported. All data will be analyzed at the end of the study. The primary analysis will be performed by the intention-to-treat approach. Everyone who begins the treatment is part of the study whether he or she completes the study or not. Additional per-protocol analysis may also be performed on subjects who complete the entire clinical trial according to the protocol. The most appropriate method of handling missing values will be chosen based on the trial's goals, endpoints and context.

The analysis of demographic, medical history, and efficacy variables will be based on all patients who receive at least one treatment and biopsies. The analysis of safety data will be based on all patients who receive at least one treatment.

## 2.16.4 Analysis of Demographic and Medical History Variables

Summaries will be prepared for all important demographic and medical history variables. For quantitative variables summaries will include the sample size, mean, median, standard deviation, minimum, and maximum. For these variables the treatment groups will be compared using either a t-test or a Wilcoxon Rank Sum test, as appropriate. For categorical variables the summaries will include the sample size and the number and percent of patients for each outcome. For these variables, the treatment groups will be compared using Fisher's Exact test. Statistical significance will be declared if the two-sided p-value is < 0.05.

## 2.16.5 Analysis of Efficacy Variables

Analysis of histological results will use biopsies from the control areas with normal skin subcutaneous adipose tissue structures and no indication of changes to be compared against the biopsies from the from the treatment areas.

## 2.16.6 Analysis of Safety Variables

Safety will be assessed through the degree of pain/discomfort related to the procedure (universal pain scale) and the collection of Adverse Events throughout the course of the study. For each treatment group these variables will be summarized. Ultrasound measurements and temperature monitoring are optional assessments and will be used for safety purposes only. The summaries will include the number and percent of patients for each outcome. No statistical comparisons will be performed for any of these variables.

#### 3.0 RISK ANALYSIS AND MANAGEMENT

## 3.1 Risk Determination

This device used in this study does not meet the FDA definition for a Significant Risk Device study per 21 CFR 812.3(m). Therefore, the Sponsor determines this is a non-significant risk device study.



\_\_\_\_\_\_

Significant risk device means an investigational device that:

- (1) Is intended as an implant and presents a potential for serious risk to the health, safety, or welfare of a subject;
- (2) Is purported or represented to be for a use in supporting or sustaining human life and presents a potential for serious risk to the health, safety, or welfare of a subject;
- (3) Is for a use of substantial importance in diagnosing, curing, mitigating, or treating disease, or otherwise preventing impairment of human health and presents a potential for serious risk to the health, safety, or welfare of a subject; or
- (4) Otherwise presents a potential for serious risk to the health, safety, or welfare of a subject.

## 3.2 Risk Management

The Investigators in this clinical trial have been invited to participate based on his/her previous experience with the use of the system and/or similar systems and industry experience. Experience with treatments is the most critical element for managing subject risk in this trial.

In addition, as with any study, there is a risk of bias. To minimize/avoid bias, objective evaluation methods (e.g. histology) will be used in conjunction with subjective evaluation methods.. The value of the compensation to the clinical investigator for conducting the study is not influenced by the study outcome. If photographic results are listed as the primary objective, they are to be evaluated by blinded evaluators who did not partake in the study. If information concerning investigator assessment of improvement or investigator satisfaction is collected, then it is not listed as an objective for the study.

All other known risks will be disclosed to the subject via the informed consent process. Since this is an elective procedure and subjects are volunteers, it can be assumed that signing the informed consent form is indicative of agreement to accept the risks involved.

Risks to subjects who participate in the study are the same as those for subjects undergoing similar noninvasive lipolysis treatment(s). It is possible to have an adverse reaction to treatment with the TempSure device . There may also be some unknown side effects.

## 3.3 Risk Analysis

## CONTEXT OF THE PROPOSED INVESTIGATION:

Radiofrequency (RF) technology is commonly used in surgery, non-invasive treatments and aesthetic applications. RF technology is a safe method for non-ablative (a non-wounding device treatment which heats underlying skin) treatment, because energy can be precisely delivered through the skin to the subcutaneous adipose tissue beneath without damaging the epidermis.

According to published data, the elevation of tissue temperature between 42°C to 47°C can affect the cellular matrix of the adipose tissue creating injury to the adipocytes and prompt an inflammatory response. Gradually, the treated adipocytes will be removed by the human body through the inflammatory clearing process which may take weeks to months. The regeneration of adipose tissue is very slow (over years) and the total volume of the fat in treatment area will decrease due to the loss of adipocytes.

## ASSESSMENT OF RISKS OF THE PROPOSED INVESTIGATION:

There are two risks identified with the TempSure® device used in this study. The first risk identified is the lack of clinical data providing evidence of effectiveness of Firm handpieces for the treatment of lipolysis. Parameters need to be further investigated to be optimized for efficacious results. The second risk identified is the safety of treatment with the TempSure® Firm handpieces. Since the TempSure® Firm handpieces have not been cleared for use for lipolysis and has limited safety data for this indication, optimizing the safety profile is necessary.

The risk identified with the overall clinical investigation is the integrity of data collected.

There are multiple clinical mitigation strategies for the risks identified. Proper training on the device and protocol will be performed. Data from prior investigations will be utilized to minimize side effects and optimize treatment outcomes. Monitoring of the study will be implemented to minimize subject and data risks.

ASSESSMENT OF BENEFITS OF THE PROPOSED INVESTIGATION:



The subject may or may not have a reduction in unwanted fat.

#### CONSIDERATION OF PATIENT PREFERENCE INFORMATION:

Many physicians support the use of radiofrequency devices for non-invasive cosmetic treatments based on current patient satisfaction. s with approved radiofrequency devices. However, there is still a level of interest in novel technologies that effectively reduce fat, potentially eliminating the need for invasive treatments for fat reduction.

#### ASSESSMENT OF UNCERTAINTY:

There is uncertainty of efficacy of treatment when TempSure® Firm is used for the treatment of unwanted fat.

#### CONCLUSION:

The TempSure® Firm handpieces used in this study have not been FDA cleared for use for the treatment of wanted fat (lipolysis) but pose no more risk than the currently cleared indications for use.

A previous safety study, CYN18-RF-TISSUE-RD, was conducted using excised human abdominoplasty tissue to test various radiofrequency parameters with the 60mm handpiece. Additional safety studies, CYN19-TS-ABDOM and CYN20-FIRM-HISTO, were conducted using patients scheduled for an abdominoplasty surgery to use in-vivo tissue to test various radiofrequency parameters with the 60mm handpiece. CYN19-TS-ABDOM used thermal measurements of treatment zones were collected to evaluate the depth of penetration and effects on human tissue. CYN20-FIRM-HISTO use biopsies to analyze histological response.

Studies CYN17-RF-CLINIC and CYN19-TS-ENVI-ABD collected safety and efficacy data using the 25mm, 30mm, and 60mm handpieces on various body areas, including the abdomen and flanks.

Patient population to be enrolled in this clinical study:

Total anticipated population: 12 Subjects Age Range years old: 18 – 55 years old

Gender: Male or Female

Condition: Unwanted fat on abdomen and scheduled for abdominoplasty surgery

## 4.0 DEVICE DESCRIPTION AND SPECIFICATIONS

The TempSure® device used in this study is currently cleared by the U.S. Food and Drug Administration (the FDA). The TempSure® device most recent 510(k) clearance under K200241 on March 25, 2020 is for:

- The 10mm, 15mm, and 20mm TempSure Envi handpieces are indicated for non-ablative treatment of mild to moderate facial wrinkles and rhytids.
- The 18mm, 25mm, 30mm, 60mm Smart Handpieces and FlexSure™ applicators provide heating for the purpose of elevating tissue temperature for selected medical conditions such as temporary relief of pain, muscle spasms, and increase in local circulation.
- The Massage device is intended to provide a temporary reduction in the appearance of cellulite.

The following surgical modes are applicable to the generator:

- Coagulation/Hemostasis: Using the surgical handpieces and accessories, general surgical procedures including urologic, thoracic, plastic, reconstructive, and gynecological procedures where electrosurgical coagulation of tissue is performed.
- Cutting: snoring. submucosal palatal shrinkage, traditional uvulopalatoplasty (RAUP), myringotomy with effective hemorrhage control, epistaxis treatment, turbinate shrinkage, skin incisions, biopsy, cysts, abscesses, tumors, cosmetic repairs, development of skin flaps, skin tags and blepharoplasty.
- Blended Cutting and Coagulation: snoring, submucosal palatal shrinkage, traditional uvulopalatoplasty (RAUP), myringotomy with effective hemorrhage control, epistaxis treatment, turbinate shrinkage, skin tags, papilloma keloids, keratosis, verrucae, basal cell carcinoma, nevi, fistulas, epithelidma, cosmetic repairs, cysts, abscesses, and development of skin flaps.



- Fulguration: basal cell carcinoma, papilloma, cyst destruction, tumors, verrucae, hemostasis.
- Bipolar: pinpoint precise coagulation, pinpoint hemostasis in any field (wet or dry). Snoring, submucosal palatal, shrinkage, traditional uvulopalatoplasty (RAUP), myringotomy with effective hemorrhage control, epistaxis treatment and turbinate shrinkage

The TempSure® device is considered investigational because TempSure® Firm handpieces used in this study are not cleared for use for lipolysis.

Changes to the TempSure® device are not anticipated during the investigation.

The TempSure® Device Specifications are:

| The Tempoures I | perice specifications are. |
|---|---|
| Surgical Connector | 1 surgical monopolar port |
| Neutral Connector | One universal neutral connector compatible with Cynosure neutral |
| | electrodes |
| Smart Handpiece | One 4-pin circular connector for both RF energy delivery and |
| Connectors | temperature sensing (monopolar) |
| Modes of | Select the Smart Handpiece or Surgical mode of operation |
| Operation | |
| Maximum Power | Temperature-Sensing Handpieces |
| | <ul> <li>▲ 10mm, 15mm, and 20mm handpieces have a maximum GUI setting of 70, which provides output power of 120 Watts (+/- 20%).</li> <li>▲ 18mm handpiece has a maximum GUI setting of 25, which provides output power of 25 Watts (+/-20%).</li> <li>▲ 25mm and 30mm handpieces have a maximum GUI setting of 80, which provides output power of 165Watts (+/- 20%).</li> <li>▲ 60mm handpieces have a maximum GUI setting of 100, which provides output power of 300 Watts (+/- 20%).</li> <li>▲ FlexSure applicators are controlled by setting the temperature. During treatment, power can reach a maximum output of 300 Watts (+/- 20%).</li> </ul> |
| | Ensuring that the neutral pad recommended for use with the 60mm handpiece and flexible applicator has sufficient current carrying capacity so as to assure that there is no unacceptable temperature rise under the pad is an essential performance of the TempSure platform. |

The TempSure® device Operator Manual: Attachment I

The TempSure® consumables are: Handpieces, NEM Pads, Gel

#### MONITORING PROCEDURES 5.0

The Sponsor Standard Operating Procedure (SOP) for monitoring the investigative site will be followed. The sponsor will train the site following sponsor SOP's and may be present at initiation of treatment. The sponsor will also monitor the site periodically. The Investigator/Institution will permit trial-related monitoring, audits, IRB/IEC review, and regulatory inspections by providing direct access to source documents. The sponsor may request intermediate data following each visit to evaluate treatment progress. Case Report Forms will be reviewed for current data and Regulatory Binders will also be reviewed for correct documents. The sponsor will collect data at the end of the follow up period. The sponsor will list the study on clinicaltrials.gov as required by FDA regulations.



The monitoring plan for this study is outlined in the Cynosure Monitoring Plan.

#### ASSIGNED CLINICAL RESEARCH MONITOR:

Monitor #1

Name: Kristy Luis

Institution: Cynosure, LLC

Address: 5 Carlisle Rd. Westford, Ma

## 6.0 LABELING

Sample labeling will follow FDA regulations and the sponsor standard operating procedure. If applicable the TempSure® device label will include, (in accordance with 801.1):

Statement: "CAUTION--Investigational device. Limited by Federal (or United States) law to investigational use."

Additionally, the label or other labeling will describe all relevant contraindications, hazards, adverse effects, interfering substances or devices, warnings, and precautions.

## 7.0 CONSENT MATERIALS

Forms and informational materials which are provided to the subject during the informed consent process are listed below:

| Form/Informational Material Description |
|-----------------------------------------|
| Pre and Post Treatment Instructions |
| Informed Consent Form |
| Universal Pain Assessment Tool |

## 8.0 INSTITUTIONAL REVIEW BOARD INFORMATION

This protocol, informed consent forms, and any amendments to the protocol will be reviewed by the appropriate Institutional Review Board prior to initiation. The study will not be initiated without the approval from the Institutional Review Board. Any action taken by any IRB will be recorded in the study file.

## **IRB Contact Information:**

IRB Name: Allendale Investigational Review Board

IRB Chairperson: Robert Staab

IRB Address: 30 Neck Rd. Old Lyme, CT 06371

Phone: 860-434-5872 Fax: 860-434-5892 Email: Rta1ali1@aol.com

#### 9.0 OTHER INSTITUTIONS

If a part of the study is conducted by an institution that has not previously been identified within the Investigational plan each institution's contact information will be documented below;

No other institutions will be part of this study.

## 10.0 ADDITIONAL RECORDS AND REPORTS

Additional records and reports will be maintained on the investigation in addition to those prescribed in 21 CFR 812.25 sub-part G.



## **Additional Records and Reports:**

| Report | Submit To | Description/Constraints |
|---|---|---|
| N/A | N/A | This is a non-IDE study; no additional records or reports will be maintained. |

## 11.0 PREGNANCY

Females may not participate in this study if they are pregnant, breastfeeding, were pregnant within the last three months or are planning a pregnancy during the study.

If the subject thinks they have become pregnant during the study, they must inform the Investigator immediately. If she becomes pregnant or thinks that she may be pregnant, she will be removed from the study and will be asked to perform a final evaluation similar to that of the final follow-up visit. The Investigator may request to track the pregnancy and will report the pregnancy to the Sponsor.

#### 12.0 SUBJECT WITHDRAWAL

The subject is free to withdraw from this study at any time. The subject must inform the Investigator immediately if they intend to withdraw. To terminate the subject's participation in this study, they must contact the Investigator at the contact information listed on page one of the informed consent form. They will be asked to come to the study clinic or Investigators office to complete a final follow up visit and may be asked to perform end of study procedures. Their decision to participate in this study or to withdraw from this study will not influence the availability of their future medical care and will involve no penalty or loss of benefits to which they are otherwise entitled.

The Investigator in charge of the study can remove the subject from this study without their consent for any reason, including, but not limited to:

- a) His/her judgment that any condition or circumstance may jeopardize their welfare or the integrity of the study.
- b) Their failure to follow the instructions of the Investigator(s).
- c) If the study is stopped by the sponsor and/or Investigators participating in the study prior to completion.

Data collected prior to withdrawal will be used in data analysis but after withdrawal no further data will be collected.

## 13.0 PHOTOGRAPHY

Standardized will be taken of the treatment area. Photographs will be taken with an appropriate high-resolution digital camera. Camera settings (lighting, distance, background, polarization, etc.) will be reproduced at each visit, so that photographs are suitable for comparison. Photographs will be taken of the treatment area for study purposes. If the subject does not wish to have their photographs taken, they cannot be in the study.

#### 14.0 ADVERSE REACTIONS DEFINITIONS AND REPORTING REQUIREMENTS

All adverse events that occur, starting from the time of the first treatment, will be recorded in the source documents and Case Report Forms (CRF).

Adverse Events (AE) occurring will be captured and followed until the condition resolves, stabilizes, is otherwise explained, or the subject is lost to follow-up. Subjects will be instructed that they may contact the Investigator at any time throughout the course of the study.



\_\_\_\_\_\_

The Investigator and/or designated study staff will review each event and assess its relationship to the study device (not related, unlikely, possible, probable, and highly probable). The following definitions will be used for rating relationship to the TempSure® Firm treatments:

- Not related The event is clearly related to other factors such as the subject's clinical state, therapeutic interventions, or concomitant medications administered to the subject.
- Unlikely The event was most likely produced by other factors such as the subject's clinical state, therapeutic interventions, or a concomitant medication administered to the subject; and does not follow a known response pattern to the investigational product.
- Possible The event follows a reasonable temporal sequence from the time of investigational product
  administration; and/or follows a known response pattern to the study sampling sessions; but could have been
  produced by other factors such as the subject's clinical state, therapeutic interventions, or concomitant
  medications administered to the subject.
- Probable The event follows a reasonable temporal sequence from the time of investigational product
  administration; and follows a known response pattern to the investigational product; and cannot be reasonably
  explained by other factors such as the subject's clinical state, therapeutic interventions, or concomitant
  medications administered to the subject.
- Highly Probable The event follows a reasonable temporal sequence from the time of investigational product administration; and follows a known response pattern to the investigational product; and cannot be reasonably explained by other factors such as the subject's clinical state, therapeutic interventions, or concomitant medications administered to the subject; and either occurs immediately following investigational product administration, or improves on stopping the investigational product, or reappears on repeat exposure, or there is a positive reaction at the application site.

Each adverse event reported will be graded on a 3-point severity. Using the following definitions for rating severity will be used:

- Mild easily tolerated, causing minimal discomfort, and not interfering with normal everyday activities.
- Moderate sufficiently discomforting and may interfere with normal everyday activities.
- Severe incapacitating and/or preventing normal everyday activities.

A Serious Adverse Event (SAE) is any adverse device experience that results in any of the following outcomes: death, a life-threatening adverse device experience, in-patient hospitalization or prolongation of hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. Important medical events that may or may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse device experience when, based upon appropriate medical judgment, they may jeopardize the subject or subject may require medical or surgical intervention to prevent one of the outcomes listed in this definition

If any of the above adverse events are serious as defined by the FDA Code of Federal Regulations (CFR), Title 21, special procedures will be followed. All serious adverse events will be reported within 24 hours of acknowledgment to the Sponsor whether or not the serious events are deemed sampling session-related. All serious event reporting will adhere to 21 CFR part 812 and the IRB will be notified accordingly.

The SAE information will be entered into the database and a desk copy of the complete SAE report will be submitted to the study file.

Adverse events, whether serious or non-serious, will be followed until the condition is resolved, stabilized, otherwise explained or the subject is lost to follow-up. Adverse events will be captured throughout the study and where appropriate, medical tests and examinations will be performed to document the resolution of event(s). Outcomes may be classified as resolved, improved, unchanged, worse, fatal, unknown or lost to follow-up. Following the resolution of any study-associated adverse events there will be no further adverse event reports for that subject.

| Reporting Adverse Events: |
|---------------------------|



| Report | Submit To | Description/Constraints |
|---|---|---|
| Adverse Events,<br>Unanticipated<br>Adverse Device<br>Effect | IRB<br>and<br>Sponsor | If an unforeseen complication is determined to be an unanticipated adverse device effect, the investigator's report must be submitted within 10 working days after the investigator first learns of the effect. |
| Serious Adverse<br>Events | IRB<br>and<br>Sponsor | The sponsor must be notified within 24 hours of serious adverse events. The IRB must be notified within 10 working days of serious adverse events as defined by FDA guidelines. |

#### 15.0 PROTOCOL DEVIATIONS

All requests for protocol deviations by the Investigator must be communicated to the sponsor in writing and if accepted by the Sponsor must be approved by the IRB. If a deviation occurs, the Investigator must inform the Sponsor as soon as possible. The Sponsor will notify the IRB in accordance with IRB specific policies.

#### 16.0 CONFIDENTIALITY AND DISCLOSURE OF MEDICAL INFORMATION

As part of this study the Investigator and the team at the research facility will keep records of subject participation in the study. These study records will include personal information that the subjects provide including age, sex, etc., the results of the study, information about response to treatments, photographs taken during the study and other medical information relating to participation in the study.

Under federal law the study records cannot be used or disclosed by the Investigator for research purposes unless subjects sign the informed consent authorization.

Some or all of the test results, photographs and other information will be reported to Cynosure, Inc. the manufacturer of the test device (Sponsor), and consultants that are helping conduct the study. The Sponsor and its consultants will analyze and evaluate these results and information and may report them to the U.S. Food Administration and the FDA, Institutional Review Board or other regulatory agencies in the United States and/or foreign countries. The subject's study records will be assigned a code number by the study team and they will ordinarily not be identified by name in the study records that are sent to the Sponsor and its consultants. However, The Sponsor, the Institutional Review Board and its consultants will have the right to see the complete study records, including the subject's name, and might choose to do so. If reports or articles are written about the study, the subject will not be identified by name in them however your study information and photographs may be used.

The research facility will review and use the study records only for purposes of this study. They will keep the subject's identity confidential and, except for the disclosures described above, will not disclose the study records to other parties unless disclosure is required by law. Once the research facility discloses information in the study records, photographs or medical records to the Sponsor or its consultants, the information will no longer be protected by federal law. Because of the need to release information to these parties, absolute confidentiality cannot be guaranteed. However, the Sponsor and its consultants will only use information for purposes of the study and will not disclose your study records to parties other than; the FDA or other regulatory agencies in the United States and/or foreign countries, unless disclosure is required by law. If reports or articles are written about the study, subjects will not be identified by name in them however, subject study information and photographs may be used.

Study records will be kept at the research facility according to applicable regulations and policies and may be kept indefinitely following the completion of the study. Subjects will not have the right to review their records while the research is in progress. However, they will be able to review their records after the research has been completed.

## 17.0 CLINICAL RESEARCH CONDUCT



\_\_\_\_\_\_

The study will be conducted in accordance with the protocol, International Conference on Harmonization (ICH) GCP guidelines, applicable regulations and guidelines governing clinical study conduct and ethical principles that have their origin in the Declaration of Helsinki. The investigator must ensure that the study is conducted in accordance with the provisions as stated in the FDA regulations and complies with the applicable local or regional regulatory requirements. The investigator will adhere to standard COVID-19 procedures as recommended by federal and state guidelines.

## 18.0 REPORTING FOR THE STUDY

A study summary report will be generated. It will include a description of the clinical conduct of the study and results.

## **Study Summary Reporting:**

| Report | Submit To | Description/Constraints |
|---|---|---|
| Deviation<br>from<br>Investigational<br>Plan | IRB<br>and<br>Sponsor | A deviation performed in an emergency to protect the life or physical well-being of a patient necessitates notification of the IRB and sponsor. The investigator's report must be submitted within 5 working days after the emergency occurred. Deviations in a non-emergency situation require notification to Sponsor prior to implementation |
| Failure to<br>Obtain<br>Informed<br>Consent | IRB<br>and<br>Sponsor | The investigator must make notification within 5 working days after device use, using the Protocol Deviation CRF. The report must include a brief description of the circumstances justifying the failure to obtain informed consent. |
| Final Report | IRB<br>and<br>Sponsor | The investigator must submit a final report within 3 months after termination or completion of the investigation. |
| Withdrawal of IRB approval | Sponsor | The investigator must report a withdrawal of the reviewing IRB approval within <u>5 working days</u> . |
| Progress<br>Report | IRB, Monitor<br>and<br>Sponsor | The investigator must submit progress reports at regular intervals, and as required by the IRB, but in no event less than annually. |

## 19.0 DISCLOSURE

The Principal Investigators, Cynosure employees and consultants have signed confidentiality agreements with the Sponsor. The confidentiality agreement ensures that all information provided to the Investigator or Data Management and Statistics departments working with the study and information obtained during the course of the study will be regarded as confidential.

## 20.0 RESPONSIBILITY OF THE INVESTIGATOR

The Investigator is responsible for ensuring the clinical study is performed in accordance with the International Conference on Harmonization (ICH), Good Clinical Practice (GCP) guidance E6, FDA Good Clinical Practice Regulations, Declaration of Helsinki (DoH) and the Health Human Service (HHS) Belmont Study. The Sponsor will comply with Financial Disclosure Rules based on pertinent financial information provided by each Investigator.

## 21.0 PROCEDURE FOR AMMENDMENTS TO PROTOCOL



Any amendment to this study will be discussed by the Investigator and the Sponsor. If agreement is reached concerning the need for modification, this will be made in a formal amendment to the protocol. With the exception of a medical emergency, deviations from this protocol will not be permitted without prior approval from the Sponsor.

All revisions and/or amendments to the protocol must be approved in writing by the appropriate Institutional Review Board.

## 22.0 TERMINATION OF STUDY

The Sponsor reserves the right to discontinue this study for administrative reasons at any time. The Investigator reserves the right to discontinue the study for safety reasons at any time in collaboration with the Sponsor.

#### 23.0 DATA SECURITY

To ensure the privacy and confidentiality of data for this protocol, the data will be stored on a restricted access private company server. Access to the project directory containing the data will be limited to the Investigators and research staff. Information about data security awareness is promoted through user training and education, supplemented by policies and procedures. Password protection will be used for all transactions that allow viewing, editing, and analysis of data, or that provide access to data fields derived from the original source documents.

## 24.0 REPORT OF PRIOR INVESTIGATIONS

The report of prior investigations or predicates are:

| Protocol | Device | IRB Name | Determination | Initial IRB<br>Approval Date |
|---|---|---|---|---|
| CYN17-RF-<br>CLINIC | TempSure/Pelleve | Allendale<br>Investigational<br>Review Board | Meets the criteria for exemption<br>from IDE regulations, non-<br>significant risk | 01/12/2017 |
| CYN18-RF-<br>TISSUE-RD | TempSure/<br>Radiofrequency<br>Devices | Allendale<br>Investigational<br>Review Board | Meets the criteria for exemption<br>from IDE regulations, non-<br>significant risk | 08/15/2018 |
| CYN19-TS-<br>ABDOM | TempSure | Allendale<br>Investigational<br>Review Board | Meets the criteria for exemption<br>from IDE regulations, non-<br>significant risk | 04/11/2019 |
| CYN19-TS-<br>ENVI-ABD | TempSure | New England IRB | Meets the criteria for exemption<br>from IDE regulations, non-<br>significant risk | 03/25/2019 |
| CYN20-FIRM-<br>HISTO | TempSure | Allendale<br>Investigational<br>Review Board | Meets the criteria for exemption<br>from IDE regulations, non-<br>significant risk | 7/2/2020 |



## APPENDIX A: Protocol Revisions Tracker

| Version<br>Date | Editor | Description |
|-----------------|-------------|----------------|
| March 5, 2020 | Kristy Luis | IRB Submission |



Appendix B

## UNIVERSAL PAIN ASSESSMENT TOOL

This pain assessment tool is intended to help patient care providers assess pain according to individual patient needs. Explain and use 0-10 Scale for patient self-assessment. Use the faces or behavioral observations to interpret expressed pain when patient cannot communicate his/her pain intensity.



REFERENCES



i Sherber, N. S., MD FAAD. (2018). The Millennial Mindset. *Journal of Drugs in Dermatology*, 17(12), 1340-1342.

ii Elsaie, M. (2009). Cutaneous Remodeling and Photorejuvenation Using Radiofrequency Devices. *Indian Journal of Dermatology*, *54*(3), 201. doi:10.4103/0019-5154.55625

<sup>&</sup>lt;sup>3</sup> American Society of Plastic Surgeons. (2019) Plastic Surgery Statics Report. Available at <a href="https://www.plasticsurgery.org/documents/News/Statistics/2019/plastic-surgery-statistics-full-report-2019.pdf">https://www.plasticsurgery.org/documents/News/Statistics/2019/plastic-surgery-statistics-full-report-2019.pdf</a>.

<sup>&</sup>lt;sup>4</sup> Centers for Disease Control and Prevention. (2020) Adult Obesity Facts. Available at <a href="https://www.cdc.gov/obesity/data/adult.html">https://www.cdc.gov/obesity/data/adult.html</a>.

<sup>&</sup>lt;sup>v</sup> Walfre Franco, et al. (2010) Hyperthermic Injury to Adipocyte Cells By Selective Heating of Subcutaneous Fat With A Novel Radiofrequency Device: Feasibility Studies. *Lasers in Surgery Medicine*. 42:361-370. DOI 10.1002/lsm.20925.

vi Katz, B., Doherty, S. (2017) Safety and Efficacy of a Noninvasive 1,064-nm Diode Laser for Fat Reduction of the Flanks. *American Society for Dermatologic Surgery, Inc.* ISSN: 1076-0512 Dermatol Surg 2017;0:1–9. DOI: 10.1097/DSS.000000000001298